CLINICAL TRIAL: NCT05149677
Title: The Effect of Music Therapy on Labour Pain, Anxiety, and Analgesia Requirement in Primiparous Patients A Randomized Controlled Clinical Trial
Brief Title: The Effect of Music Therapy on Labour Pain, Anxiety, and Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC MN178 20/21
Record Dates: First submitted 2021-11-08; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-10

CONDITIONS: Labor Pain
Keywords: pain; anxiety; labour; primiparous; music; therapy
MeSH Terms: conditions — Labor Pain; Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care for labor pain (No Intervention): Standard of Care of Care for labor pain
- Music therapy intervention + Standard of Care for labor pain (Experimental): Music therapy intervention + Standard of Care for labor pain
  Interventions: Behavioral: Music therapy

INTERVENTIONS:
Behavioral: Music therapy — Music therapy intervention + Standard of Care for labor pain
  Arms: Music therapy intervention + Standard of Care for labor pain

SUMMARY:
Labour pain is the result of complex and subjective interactions of multiple physiologic and psychosocial factors on a woman's interpretation of labour stimuli. It is an integral part of the labour process, often associated with anxiety and being subjective, affects each woman's experience of the birthing process in differing ways.

This will be a randomized clinical trial, involving primiparous women presenting to the University Hospital of the West Indies (UHWI) for labour and delivery. Primiparous, term women in labour will be eligible and randomized in a 1:1 ratio to receive music plus standard of care during labour and standard care without music therapy.

The primary outcome of this study will be to determine whether music therapy is an effective adjunct or alternative to pharmacological therapies for pain and anxiety management in labour. The secondary outcome would be to assess the effect of music on labour duration, operative delivery rates, abnormal foetal heart rate patterns and APGAR scores. Approximately 260 primigravida women would be recruited and invited to participate in this randomized clinical trial over an eight-month period.

DETAILED DESCRIPTION:
The Cambridge dictionary describes pain as a feeling of physical suffering caused by injury and illnesses. This physical suffering is a subjective, natural, and inevitable process associated with labour that is understandably, a most feared aspect of pregnancy for expectant mothers. A woman's birthing experience is influenced by her social environment and how she contextualizes the idea of pain as purposeful and productive versus threatening, the latter of which could result in a more negative pain response. Historically prior to the 18th century, natural methods were the only options for pain relief for women in labour. These included various breathing techniques and positioning, massage techniques and herbal mixtures. There is an increasing movement back to the historical practices of traditional and non- pharmacological pain relief during labour, and research in these techniques is needed to prove clinical effectiveness. According to the World Health Organisation (WHO) recommendations: intrapartum care for a positive childbirth experience- " Most women desire some form of pain relief during labour, and qualitative evidence indicates that relaxation techniques can reduce labour discomfort, relieve pain and enhance the maternal birth experience."

One of the most used pharmacological agents during labour is meperidine hydrochloride (Pethidine®) as it is readily available with a higher level of administrator comfort than other agents. Overuse of pharmacological interventions can lead to increased maternal and neonatal morbidity, reduced local supply of pharmacological agents and even financial strain on low resource institutions. Patients with a low pain threshold in early labour due to anxiety and fear may also request analgesia in the latent phase which can result in the inability to receive repeated doses early in the active phase due to dosing frequency guidelines. This can then result in maternal distress and poor labour outcomes when the additive effect of labour progression, results in more severe pain. Meperidine hydrochloride has been shown to offer variable pain control with a more sedation than analgesic effect, hence adjunctive therapy with music may prove beneficial for its potential additive analgesic effect. Meperidine hydrochloride's use has also been found to be associated with increased rate of augmentation in labour, increased operative deliveries, and adverse maternal effects such as nausea, vomiting and dizziness and also a linkage to neonatal respiratory depression & APGAR scores < 7 and acidosis [umbilical artery potential of Hydrogen (pH) <7.12] have been noted.

The United Nation (UN) Global Strategy for Women's, Children's and Adolescents' Health seeks to ensure that not only do women survive childbirth complications if they arise, but also that they thrive and reach their full potential for health and life. To facilitate safe labour and childbirth, attention must be given to the management of the psychological and emotional needs of women. Anxiety of the labour process is frequently seen in mothers presenting for delivery. This is shown to be more common in primiparous women especially if they have not received antenatal counselling on what to expect in labour(9). Studies have shown that anxiety can stimulate the sympathetic nervous system, releasing excessive stress hormones such as cortisol and adrenaline contributing to dysfunctional uterine contractility and labour dystocia. Music therapy has been shown to be an effective, inexpensive, safe and non-invasive intervention for patients undergoing many non-obstetric procedures such as decreased pain and anxiety during bone marrow biopsy and aspiration and nasal bone fracture reduction as well as decreased anxiety and propofol (Diprivan®) consumption during colonoscopy/endoscopy.

With more women exploring the option of physiological birthing techniques ("Natural Birthing Techniques"), an approach to labour and birth that normalizes the strength and physiology of the woman and foetus and refrains from external intervention unless there is potential compromise to mother or foetus, music therapy may offer a natural alternative to pharmacological approaches to pain relief that are the standard of care in may labour and delivery suites.

Music can have a direct impact on the perception of pain by activating the gate-control theory of pain which attacks both cognitive and physiological factors associated with pain. The gate theory works on the idea that there is a gateway in the dorsal horn of the spinal cord that manages the perception of pain via opening and closing of this gate. Pain sensation is carried via small neural fibres that pass this gate in route to the brain for interpretation. Music can close this gateway by stimulating a large number of neurological fibres some of which would have been activated for a pain response if available, and hence no transmission of pain sensation in response to stimulation. Music can also serve as a distraction mechanism improving general mood and hence decreasing negative pain perception.

Music during labour is perceived by the right hemisphere of the brain and can result in the release of endorphins which provide analgesia by binding to opioid receptors at pre and post synaptic nerve terminals. This binding results in the inhibition of substance P an important protein involved in the transmission of pain. Studies show that decreased levels of serum cortisol and the release of neural system of reward hormones such as dopamine is linked to the anxiety reducing effect of music therapy.

In a study performed by Buglione et al., pain level during active phase of labour was 8.8 ± 0.9 in music group and, 9.8 ± 0.3 in control group [Mean Difference (MD) - 1.00 point, 95%, Chloride (Cl) - 1.48 to - 0.52; P <0.01]. Music during labour and delivery was also associated with decreased pain 1h postpartum as well as decreased anxiety levels during the active phase, second stage and 1hour postpartum. This study was however studied in a small population of 30 Italian women; hence generalizability of findings is uncertain. A meta-analysis and systematic review of studies published between 2003 and June 2018 showed significant differences in Visual Analog pain scale (VAS) scores in favour of music therapy in the intensity of latent phase of labour pain (MD: -0.73; 95% Cl -0.99, -0.48); in the active phase (MD: -0.68; 95% Cl -0.92, -0.44) in its entirety or during the first phase (MD: -1.71; 95% Cl -2.65, -0.77) and second hour postintervention (MD: -2.90; 95% Cl -3.79, -2.01). In terms of anxiety, Santiváñez-Acosta et al evaluated three studies which revealed significant differences in anxiety level in the latent phase (MD: -0.74; 95% Cl -1.00, -0.48) and active phase of labour (MD: -0.76; 95% Cl -0.88, -0.64).

ELIGIBILITY:
Inclusion Criteria:

* Women attending the UHWI antenatal clinic (General antenatal clinic or departmental antenatal clinic)
* Primiparous
* Age 18 years and over
* ≥ 37weeks pregnancy
* Singleton Foetus
* Consent to participate in study

Exclusion Criteria:

* Multiparous
* Preterm pregnancy
* Multiple Gestation
* Planned Caesarean Section
* Epidural Analgesia or treatment antipsychotic medication
* Comorbid illness: maternal hypertensive disorders, diabetes mellitus, evidence of intrauterine growth restriction, suspected macrosomia, premature rupture of membranes, maternal hearing difficulties, chronic pain problems, severe dysmenorrhea, foetal death in utero, known cardiovascular or another foetal anomaly
* inability to understand the visual analogue scale
* No consent to participate in study

Ages: 18 Months to 65 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — women 37 and 41 weeks of gestation in labour
Enrollment: 260 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
difference in mean pain visual pain score between standard of care group during latent phase of labor and Music therapy intervention group | Duration in hours from admission until the end of latent phase of labour
  Pain will be assessed during each 30-minute intervals following consecutive hourly observations using a self-reported visual analogue scale with range of scores from 0 to 10 with 0 indicating no pain and 10 indicating maximum pain during the latent phase of labour (cervical dilation 2-4 cm). The mean pain scores during phase will be computed for each group (music therapy group with standard of care and the standard of care group ) and their mean difference compared.
difference in mean pain visual pain score between standard of care group during active phase of labor and Music therapy intervention group | Duration in hours from start of active phase for up to 3 hours.
  Pain will be assessed during each 30-minute intervals following consecutive hourly observations for 3 hours using a self-reported visual analogue scale with range of scores from 0 to 10 with 0 indicating no pain and 10 indicating maximum pain during the latent phase of labour (cervical dilation >=5 cm). The mean pain scores during active phase will be computed for each group (music therapy group with standard of care and the standard of care group ) and their mean difference compared.
difference in pain visual pain score between standard of care group 2 hours post delivery of labor and Music therapy intervention group | At 2 hours post delivery
  Pain will be assessed at 2 hours post delivery using a self-reported visual analogue scale with range of scores from 0 to 10 with 0 indicating no pain and 10 indicating maximum pain. The pain scores at 2 hours post-delivery will be assessed for each group (music therapy group with standard of care and the standard of care group ) and their mean difference compared.
difference in duration of labour between standard of care group during active phase of labor and Music therapy intervention group | Duration in hours from admission until delivery
  The duration of latent and active phase of labour will be measured in minutes for each participant in each group (music therapy group with standard of care and the standard of care group ) and their mean computed. The difference in mean duration of labor by groups will be compared.

SECONDARY OUTCOMES:
Difference in mean APGAR score at 5 minutes post -delivery of children of mothers assigned to standard of care group and Music therapy intervention group. | At 5 minutes post delivery
  The APGAR score at 5 minutes for each infant born to mothers assigned to (music therapy group with standard of care and the standard of care group ) will be assessed and the group means computed. The difference in mean APGAR score by groups will be compared.
Difference in mean cumulative amounts of analgesia used during labor and delivery for mothers assigned to standard of care group and Music therapy intervention group. | Duration in hours from admission until delivery
  The amounts of analgesia used for each woman during labour and delivery will be recorded.The amounts of analgesia used will be converted to equianalgesic doses. The difference in mean cumulative equianalgesic amounts by groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Rattray, Principal Investigator — University Hospital of the West Indies Mona Jamaica- Maternity Delivery Unit; M Campbell-Mitchell, Principal Investigator — University Hospital of the West Indies Mona Jamaica- Maternity Delivery Unit
Locations (1):
- University of the West Indies Mona Jamaica, Kingston, Jamaica